CLINICAL TRIAL: NCT05285605
Title: Advance Provision of Postpartum Emergency Contraception and Its Effects on Reproductive Autonomy
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Other Study IDs: STU00215994
Record Dates: First submitted 2022-03-06; First posted 2022-03-17 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-03

CONDITIONS: Contraception; Contraceptive Usage; Reproductive Issues
Keywords: Emergency Contraception; Reproductive Autonomy
MeSH Terms: conditions — Contraception Behavior | interventions — ulipristal acetate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Emergency Contraceptive Group: Group of participants receiving emergency contraception in the form of 3 packages of ulipristal acetate to use at home if needed.
  Interventions: Drug: Ulipristal Acetate

INTERVENTIONS:
Drug: Ulipristal Acetate — Ulipristal acetate 30mg x 1 dose as needed for unprotected intercourse
  Other Names: Ella

SUMMARY:
This study will entail provision of ulipristal acetate (UPA) for emergency contraception (EC) in the postpartum period for patients who have not chosen to initiate a highly effective form of contraception and study the use of EC overall as well as with regards to participants' perception of reproductive autonomy. The investigators hypothesize that providing an advance supply of EC will increase use and decrease barriers to use. Additionally, the investigators hypothesize that, with thorough EC counseling, participants will develop an increased knowledge base of EC. With increased use and knowledge, the investigators hypothesize that participants will experience greater reproductive autonomy over their contraceptive decisions.

DETAILED DESCRIPTION:
This project will be a prospective observational study, using a mixed-methods design to further explore the impact of emergency contraception (EC) use on postpartum patients' feelings of reproductive autonomy. The investigators will aim to recruit 75 participants, with an expected 40-50 participants retained at 6 months, and 15-20 of those participants choosing to participate in an in-depth interview at 6 months. Participants will first be screened for eligibility on chart review. If any inclusion/exclusion criteria remain unclear in the medical record, these participants will still be approached to complete the eligibility survey if they are interested in participating in the study. All potential participants will confirm their contraceptive method prior to enrolling in the study. Participants who are undecided on their postpartum contraceptive plan will not meet inclusion criteria for the study. This is to avoid possible coercion or influence by the research study on patients' contraceptive choices.

If they choose to enroll in the study, they will undergo an informed consent and a baseline survey comprised of standard demographic questions, questions on reproductive and contraceptive history, knowledge on EC, and questions on reproductive autonomy. This survey will be designed to take ~10 minutes to complete. Participants will undergo standardized counseling on postpartum contraception. This counseling will include 1) best-practice recommendation for high-efficacy postpartum contraception, 2) recommendation for appropriate pregnancy spacing, 3) efficacy of contraceptive methods, and 4) types of EC and detailed instructions for use. They will receive a package of three doses of UPA prior to being discharged home along with educational material for EC. If participants need additional doses of EC, they would be able to call the clinic for additional doses. Participants will then complete surveys at 6 weeks, 3 months, and 6 months. In the 6-week survey, if they have used EC by that time, they will be invited to participate in a brief, 20-30 minute interview that will focus on their experience, comfort, and facilitators/barriers to their most recent EC use. In the 6-month survey, the participant will be invited to participate in an in-depth interview designed to further explore participant experiences with EC. The qualitative interview is expected to last ~1 hour and will discuss themes around EC use, acceptability, autonomy, contraceptive choice.

ELIGIBILITY:
Inclusion Criteria:

* 16-40 years of age
* English-speaking
* In a sexual relationship with possibility of pregnancy
* Delivered a live infant
* Desire to delay pregnancy for at least a year
* A patient at Northwestern University Feinberg School of Medicine Department of Obstetrics and Gynecology
* Choosing no postpartum contraceptive method or a lower efficacy method: condoms, female condoms, diaphragm/cervical cap/sponge, fertility awareness method

Exclusion Criteria:

* Allergy to UPA
* Those who have had tubal sterilization
* Those who conceived via assisted reproductive technology
* Those with inability to follow up
* Those taking drugs that interact with UPA (CYP3A4 inducers, abametapir, felbamate, fexinidazole, fusidic acid, griseofulvin, oxcarbazepine, progestins, topiramate)

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The participants recruited for this study originate from a diverse group of obstetrics clinics, including a resident-run clinic, an academic faculty low-risk obstetric clinic, an academic high-risk obstetric clinic, and a high-risk fellow-run clinic. The majority of these participants are residents of Chicago and its metro area. These clinics see patients with public and private insurances, and the population is expected to be similarly diverse to the city of Chicago.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in reproductive autonomy | Reproductive autonomy will be assessed at baseline, 6 weeks, 3 months, and 6 months.
  Uses a modified reproductive autonomy scale to measure participants' sense of reproductive autonomy. Highest score is 40 which is associated with greater reproductive autonomy and lowest score is 0.

SECONDARY OUTCOMES:
Change from baseline in knowledge around emergency contraception | Knowledge is assessed at baseline, 6 weeks, 3 months, and 6 months
  Uses a survey that measures knowledge on emergency contraception. Highest score is 18 and lowest score is 0. Higher scores are associated with increased knowledge on emergency contraception
Number of participants who use emergency contraception during study period | Throughout the study period, assessed at 6 months.
  Follow up surveys will ask participants if they have used emergency contraception and how many times. This will be compared with the total number of study participants in the study to denote the percentage of participants who used emergency contraception.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley M Turner, MD MSc, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern Medicine Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT05285605/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT05285605/ICF_001.pdf